CLINICAL TRIAL: NCT05429684
Title: Precise Targeted Therapy for Refractory HER2 Positive Advanced Breast Cancer Based on Genome Signature and Drug Sensitivity of PDO Model
Brief Title: Precise Therapy for Refractory HER2 Positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2020-006
Record Dates: First submitted 2021-12-12; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: HER2+ Breast Cancer
MeSH Terms: interventions — Trastuzumab; pertuzumab; Taxes; Albumin-Bound Paclitaxel; pyrotinib; Capecitabine; Ado-Trastuzumab Emtansine; Everolimus; palbociclib; Letrozole; spartalizumab; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A. HER2 low expression (Experimental): Phenotype was signatured by HER2 low expression.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Nab paclitaxel
- B. HER2 amplified (Experimental): Signatured by wild type HER2 amplified.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Nab paclitaxel
- C. HER2 mutation (Experimental): Signatured by HER2 mutation.
  Interventions: Drug: Pyrotinib; Drug: Capecitabine
- D. HER2 downstream mutation (Experimental): Signatured by HER2 downstream mutation of PI3KCA, TP53 or PTEN.
  Interventions: Drug: Trastuzumab; Drug: Nab paclitaxel; Drug: T-DM1; Drug: Everolimus
- E. Hormone receptor pathway activation (Experimental): Signatured by both ER and PR strongly expressed,or CCND1 amplified.
  Interventions: Drug: Trastuzumab; Drug: CDK4/6 inhibitor; Drug: AI
- F. Immune activation (Experimental): Signatured by high TMB or PD-L1 positively expressed.
  Interventions: Drug: Trastuzumab; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab (6mg/Kg, iv.drip, d1, q3w)
  Other Names: herceptin；Inetetamab
  Arms: A. HER2 low expression; B. HER2 amplified; D. HER2 downstream mutation; E. Hormone receptor pathway activation; F. Immune activation
Drug: Pertuzumab — Patuzumab (420mg iv.drip, d1,q3w)
  Other Names: Perjeta
  Arms: A. HER2 low expression; B. HER2 amplified
Drug: Nab paclitaxel — nab-paclitaxel (200mg iv.drip, d1,d8, q3w)
  Other Names: Abraxane
  Arms: A. HER2 low expression; B. HER2 amplified; D. HER2 downstream mutation
Drug: Pyrotinib — Pyroltinib (400mg po qd)
  Other Names: SHR-1258
  Arms: C. HER2 mutation
Drug: Capecitabine — Capecitabine (1250mg/m2, po, bid, d1-d14, q3w).
  Arms: C. HER2 mutation
Drug: T-DM1 — T-DM1(3.6mg/Kg, iv.drip, d1, q3w)
  Other Names: Trastuzumab Emtansine
  Arms: D. HER2 downstream mutation
Drug: Everolimus — Everolimus (4mg, po, qd)
  Other Names: RAD001
  Arms: D. HER2 downstream mutation
Drug: CDK4/6 inhibitor — Palbociclib (125mg, po, qd)
  Other Names: Palbociclib；
  Arms: E. Hormone receptor pathway activation
Drug: AI — Letrozole (2.5mg, qd).
  Other Names: Letrozole
  Arms: E. Hormone receptor pathway activation
Drug: Anti-PD-1 monoclonal antibody — Cindilimab (200mg, iv.drip, d1, q3w)
  Other Names: Sintilimab
  Arms: F. Immune activation

SUMMARY:
This is an open, prospective and interventional clinical study. Patients with advanced Human Epidermal Growth Factor Receptor 2 (HER2) positive breast cancer resistant to trastuzumab will be enrolled in the study. Histological specimens obtained from different metastatic foci of patients, are used to conduct genome-wide sequencing together with Circulating tumor DNA (ctDNA) of blood samples. Meanwhile, investigator will construct PDO model based on biopsy tissue. Patients as well as their paired Patient-derived organoids (PDO) models are divided into six groups according to genomic signatures. Each group of patients will receive the best targeted treatment scheme from the current clinical perspective, while the matched PDO model will accept a variety of potential effective schemes intervention. The future treatment plan of patients will be timely adjusted based on the tumor inhibition rate of PDO models. This study is the first time to explore the best individualized application sequence of targeted therapy for refractory HER2 positive breast cancer by combining genome sequencing with drug sensitivity test of PDO model. The results are expected to improve the prognosis of patients with advanced HER2 positive breast cancer.

DETAILED DESCRIPTION:
In previous studies, investigator found that dynamic genomics detection of metastatic foci can fully reveal the mechanism of trastuzumab resistance. Different anti-HER2 treatment strategies for different mechanisms can improve the efficacy of HER2 positive advanced breast cancer, and the PDO drug sensitivity test model of breast cancer can be prior to patients' response to the exact efficacy of specific regimens.This study aimed to explore the optimal individualized drug combination and order for patients with advanced HER2 positive breast cancer resistant to trastuzumab based on a variety of existing diagnosis and treatment methods. This is an open, prospective and interventional clinical study. Patients with advanced HER2 positive breast cancer resistant to trastuzumab will be enrolled in the study. Histological specimens obtained from different metastatic foci of patients, are used to conduct genome-wide sequencing together with ctDNA of blood samples. Meanwhile, investigator will construct PDO model based on biopsy tissue. Patients as well as their paired PDO models are divided into six groups according to genomic signatures. Each group of patients will receive the best targeted treatment scheme from the current clinical perspective, while the matched PDO model will accept a variety of potential effective schemes intervention. The future treatment plan of patients will be timely adjusted based on the tumor inhibition rate of PDO models. This study is the first time to explore the best individualized application sequence of targeted therapy for refractory HER2 positive breast cancer by combining genome sequencing with drug sensitivity test of PDO model. The results are expected to improve the prognosis of patients with advanced HER2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old;
2. Women;
3. ECOG score 0-2;
4. Locally advanced or metastatic breast cancer confirmed by histopathology;
5. Positive HER2 expression in cancer tissues (IHC 3 +, or IHC 2 + but FISH amplification);
6. Resistant to trastuzumab (including disease progression during or after withdrawal of trastuzumab);
7. There were enough specimens for immunohistochemistry, gene detection and establishment of PDO model;
8. Hematology and liver and kidney function were normal within 2 weeks before treatment;
9. Imaging examination showed measurable lesions (according to RECIST v1.1);
10. Women of childbearing age agree to contraception or take contraceptive measures;
11. Be able to understand the research program and participate voluntarily.

Exclusion Criteria:

1. Symptomatic, untreated or progressive central nervous system metastases;
2. Severe heart disease (poor cardiac function);
3. Within 5 years, there was a history of other malignant tumors other than breast cancer;
4. In this study, chemotherapy, radiotherapy, immunotherapy or surgery were performed within 3 weeks before the first treatment;
5. Patients who are pregnant or lactating, or plan to become pregnant during enrollment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to six weeks, first evaluation
  objective response rate (ORR) according to RECIST (version 1.1) of each group
PDO model inhibition rate | during the procedure
  Tumor regression rate based on the calculation of the long diameter in each group

SECONDARY OUTCOMES:
PFS1 | during the procedure
  Progress free survival (PFS) according to RECIST (version 1.1) of each group

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Doctor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jin Yang, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No